A comparison of four different treatment regimens as the first-line treatment of Helicobacter pylori in Chinese children and investigation of resistance -a multicenter study

| RESEARCH ETHICS BOARD APPROVAL | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| PROTOCOL | TITLE: | A | comparison | of | four | different | treatment | regimens | as | the |
| PROTOCOL TITLE: A comparison of four different treatment regimens as the first-line treatment of Helicobacter pylori in Chinese children and investigation | | | | | | | | | | |
| of resistance -a multicenter study | | | | | | | | | | |
| 01 10010 | | | | | | | | | | |
| | | | | | | | | | <b>a</b> " | |

PRIMARY INVESTIGATORS: Zhou Ying

PROTOCOL TYPE: ①for PhD degree② "star fund" supported by HealthCare Nutrition of Nestle

APPLICATION INSTITUTIONS: Children's Hospital of Fudan University

STARTING AND ENDING DATES: 2017. 10-2020. 10

NAME LIST OF RESEARCH ETHICS BOARD: Zhu qi-rong;; Zhou wen-hao; Xiao xian-min; Lu yi-qun; Qiu zi-long; Xing qing-he; Kan hai-dong; Qian li-ling; Shi xiao-hua; Yin yin

THE FOLLOWING ITEMS ARE COMPLETED BY RESEARCH ETHICS BOARD:

| DOCUMENTS: | (CLICK | √ | BEFORE OPINION) |
|------------|--------|---|-----------------|

(  $\checkmark$ ) protocol

 $(\sqrt{})$  application form

(  $\sqrt{\phantom{a}}$  informed and consent form

( ) relevant approvals

( ) other informations

## RESEARCH ETHICS BOARD'S OPINION (CLICK ✓ BEFORE OPINION)

 $(\sqrt{})$  approval

( ) to be re-investigated in case of supplying supplementary documents

( ) disapproval

REMARKS:

CHAIRMAN'S SIGNATURE::



2017.9.2)